CLINICAL TRIAL: NCT03959969
Title: Educational Video on Pain Management and Subsequent Opioid Use After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Sara N. Iqbal, Maternal Fetal Medicine Fellowship Program Director, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00000260
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Opioid Use, Unspecified
MeSH Terms: interventions — Standard of Care; Ibuprofen; Oxycodone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational Video Recipients (Experimental): Participants will be shown educational video on pain management after cesarean delivery on day of discharge. Upon discharge, participants will be given twenty tablets of oxycodone 5 mg by mouth every four hours as needed for pain and forty tablets of ibuprofen 600 mg by mouth every six hours as needed for pain.
  Interventions: Other: Educational video; Drug: Ibuprofen; Drug: Oxycodone
- Standard of Care Recipients (Active Comparator): Participants will be given standard of care discharge instructions for pain management on day of discharge. Upon discharge, participants will be given twenty tablets of oxycodone 5 mg by mouth every four hours as needed for pain and forty tablets of ibuprofen 600 mg by mouth every six hours as needed for pain.
  Interventions: Other: Standard of care; Drug: Ibuprofen; Drug: Oxycodone

INTERVENTIONS:
Other: Educational video — An educational video on pain management after cesarean section. The educational video was put together by two general obstetrician-gynecologists, two maternal fetal medicine specialists, and a palliative care physician.
  Arms: Educational Video Recipients
Other: Standard of care — The standard of care discharge instructions for postoperative patients after cesarean section that are provided at the institution.
  Arms: Standard of Care Recipients
Drug: Ibuprofen — Prescription given for forty tablets of ibuprofen 600 mg every 6 hours as needed for pain.
  Other Names: Advil
Drug: Oxycodone — Prescription given for twenty tablets of oxycodone 5 mg every 4 hours as needed for pain.

SUMMARY:
This is a randomized controlled trial assessing the utility of an educational video on pain management after a cesarean section to reduce opioid use. The educational video will be shown during the patient's postpartum stay and the amount of opioid and adjunct medications will be assessed in those who watched the video compared to those who received the standard of care discharge instructions without the video. Participants will be contacted 7 and 14 days after cesarean birth (post operative day number 7 and number 14) to complete a telephone survey on their overall pain management and to determine how many opioid tablets have been used.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Underwent repeat or primary C-section
* Literate in English Language

Exclusion Criteria:

* Complicated cesarean section including cesarean hysterectomy, bowel injury, bladder injury, and/or take-back
* History of opioid use disorder and/or on chronic opiates in pregnancy
* Contraindications to NSAIDS or acetaminophen

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-01-11 (Actual)

PRIMARY OUTCOMES:
Number of oxycodone tablets used fourteen days after cesarean delivery | A total of 14 days after cesarean delivery (postpartum day number 14)
  This is the total number of oxycodone tablets used by participants in each arm fourteen days after cesarean delivery (postpartum day number 14).

SECONDARY OUTCOMES:
Pain assessment score from numeric pain intensity scale at seven days after cesarean delivery | 7 days after cesarean delivery (postpartum day number 7)
  Using an universal pain assessment tool of a numeric pain intensity scale, patients will be asked their pain score seven days after cesarean delivery (postpartum day 7). The numeric pain intensity scale is 0-10, with 0 being no pain and 10 being the worst pain possible.
Adjunct medication use at seven days after cesarean delivery | 7 days after cesarean delivery (postpartum day number 7)
  This is to determine use of adjunct medications such as ibuprofen and Tylenol in the participants in both arms, seven days after cesarean delivery.
Overall pain management satisfaction using Likert scale seven days after cesarean delivery | 7 days after cesarean delivery (postpartum day number 7)
  Assessment of overall pain management satisfaction seven days after cesarean delivery (postpartum day number 7) with five point Likert scale. The Likert scale ranges from extremely satisfied with pain management to extremely dissatisfied with pain management.
Pain assessment score from numeric pain intensity scale at fourteen days after cesarean delivery | 14 days after cesarean delivery (postpartum day number 14)
  Using an universal pain assessment tool of a numeric pain intensity scale, patients will be asked their pain score fourteen days after cesarean delivery (postpartum day 14).The numeric pain intensity scale is 0-10, with 0 being no pain and 10 being the worst pain possible.
Adjunct medication use at fourteen days after cesarean delivery | 14 days after cesarean delivery (postpartum day number 14)
  This is to determine use of adjunct medications such as ibuprofen and Tylenol in the participants in both arms, fourteen days after cesarean delivery.
Overall pain management satisfaction using Likert scale fourteen days after cesarean delivery | 14 days after cesarean delivery (postpartum day number 14)
  Assessment of overall pain management satisfaction fourteen days after cesarean delivery (postpartum day number 14) with five point Likert scale. The Likert scale ranges from extremely satisfied with pain management to extremely dissatisfied with pain management.
Total number of oxycodone tablets used inpatient | 3 days
  Total oxycodone tablets used during patient's inpatient stay after cesarean delivery.
Number of oxycodone tablets used seven days after cesarean delivery | 7 days after cesarean delivery (postpartum day number 7)
  This is the total number of oxycodone tablets used by participants in each arm seven days after cesarean delivery (postpartum day number 7).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Iqbal, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prabhu M, McQuaid-Hanson E, Hopp S, Burns SM, Leffert LR, Landau R, Lauffenburger JC, Choudhry NK, Kaimal A, Bateman BT. A Shared Decision-Making Intervention to Guide Opioid Prescribing After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):42-46. doi: 10.1097/AOG.0000000000002094. PMID 28594762
- [Background] Bateman BT, Cole NM, Maeda A, Burns SM, Houle TT, Huybrechts KF, Clancy CR, Hopp SB, Ecker JL, Ende H, Grewe K, Raposo Corradini B, Schoenfeld RE, Sankar K, Day LJ, Harris L, Booth JL, Flood P, Bauer ME, Tsen LC, Landau R, Leffert LR. Patterns of Opioid Prescription and Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):29-35. doi: 10.1097/AOG.0000000000002093. PMID 28594763
- [Background] Ismail S, Shahzad K, Shafiq F. Observational study to assess the effectiveness of postoperative pain management of patients undergoing elective cesarean section. J Anaesthesiol Clin Pharmacol. 2012 Jan;28(1):36-40. doi: 10.4103/0970-9185.92432. PMID 22345943
- [Background] ACOG Committee Opinion No. 742 Summary: Postpartum Pain Management. Obstet Gynecol. 2018 Jul;132(1):252-253. doi: 10.1097/AOG.0000000000002711. PMID 29939935
- [Derived] Mokhtari NB, Saeed H, Kawakita T, Huang JC, Iqbal SN. Educational Video on Pain Management and Subsequent Opioid Use After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2021 Aug 1;138(2):253-259. doi: 10.1097/AOG.0000000000004468. PMID 34237764